CLINICAL TRIAL: NCT06663657
Title: Effects of Cognitive Sensorimotor Exercises Versus Task Oriented Training on Balance ,Gait and Activities of Daily Living in Chronic Stroke Patients.
Brief Title: Effects of Cognitive Versus Task Oriented Training on Balance, Gait and Daily Activity in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0201
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Stroke, Ischemic; Cognitive Impairment; Balance; Distorted; ADL
Keywords: Stroke, Ischemic; Cognitive Impairment; Balance; Distorted; ADL
MeSH Terms: conditions — Ischemic Stroke; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: the patients will be randomized by lottery method and allocated into two intervention groups. Patients in group A will receive cognitive sensorimotor exercises for 30 minutes, sessions for 5 days per week for 8 weeks. Patients in group B will receive task-oriented training for 30 minutes, sessions for 5 days per week for 8 weeks. Intervention will be applied for 8 weeks it include taking reading 1st at baseline, 2nd reading at 4th week and 3rd reading at 8th week and follow up after 12 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive sensorimotor exercise group (Experimental): Patients in group A will receive cognitive sensorimotor exercises for 30 minutes, sessions for 5 days per week for 8 weeks.
  Interventions: Other: Cognitive Sensorimotor Exercises
- Task based training group (Active Comparator): Patients in group B will receive task oriented training for 30 minutes, sessions for 5 days per week for 8 weeks.
  Interventions: Other: Task Oriented Training group

INTERVENTIONS:
Other: Cognitive Sensorimotor Exercises — Patients in group A will receive cognitive sensorimotor exercises for 30 minutes, sessions for 5 days per week for 8 weeks.
  Arms: cognitive sensorimotor exercise group
Other: Task Oriented Training group — Patients in group B will receive task oriented training for 30 minutes, sessions for 5 days per week for 8 weeks.
  Arms: Task based training group

SUMMARY:
To determine effects of cognitive sensorimotor exercises versus task oriented training on balance, gait and activities of daily living in chronic stroke patients.

DETAILED DESCRIPTION:
This study will be randomized clinical trial with total of 40 participants with chronic stroke. Patients will be recruited from Riphah rehabilitation centre and National Hospital Lahore. The sampling technique will be non probability convenience sampling technique. The patients will be randomized by lottery method and allocated into two intervention groups.

Patients in group A will receive cognitive sensorimotor exercises for 30 minutes, sessions for 5 days per week for 8 weeks. Patients in group B will receive task-oriented training for 30 minutes, sessions for 5 days per week for 8 weeks. Intervention will be applied for 8 weeks it includes taking reading 1st at baseline, 2nd reading at 4th week and 3rd reading at 8th week and follow up after 12 weeks. The assessment tools used will be berg balance test for balance, Dynamic gait index for gait and Modified Barthel index to assess activities of daily livings. Data will be analysed by using SPSS 25 version.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic stroke (6 months to 2 years)
* Patients with the ability to walk independently using aids or orthotics with or without supervision.
* Ability to communicate and follow instructions.
* No problem walking due to ankle contracture.
* No sensory deficiencies of the lower extremities.
* Patients cognition level on MMSE ≥ 24

Exclusion Criteria:

* Recent injuries- Patients having musculoskeletal or surgical problems of lower extremity.
* Co-morbid conditions- Cardiovascular (uncontrolled high blood pressure, diabetes), respiratory problems like dyspnoea.
* Neurological conditions- like brain tumour, demyelinating disease, Parkinson's disease, multiple sclerosis).
* Subjects with auditory and vestibular disorders.
* Cerebellar related problems.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
The BBS (Berg Balance Scale) | 10 months
  The BBS (Berg Balance Scale) comprises 14 items aimed at evaluating balance function in older adults residing in the community. Each item is scored on a 5-point scale, ranging from 0 to 4, with a total score range of 0 to 56. Higher scores indicate better balance function. The scale exhibits robust psychometric properties, including good internal consistency (Cronbach's α = 0.92-0.98), strong interrater reliability (interclass correlation coefficient = 0.97), and favorable concurrent validity (high correlations [r = 0.91-0.95] with the PASS and the Static Balance Test).
The DGI (Dynamic Gait Index) | 10 months
  The DGI (Dynamic Gait Index) is an eight-item assessment tool designed to evaluate balance, functional mobility, and gait. Notably, the evaluation setting lacked stairs, prompting subjective patient reporting for the stair climbing item to facilitate completion of the measure. Importantly, research supports that omitting the stair component does not compromise the validity or integrity of the DGI. Each of the eight DGI items is scored on a 4-point scale, where a score of 3 indicates no gait dysfunction, 2 reflects minimal dysfunction, 1 represents moderate dysfunction, and 0 denotes severe dysfunction. The total maximum score achievable is 24. The test can be administered in approximately 10 minutes,
The Modified Barthel Index | 10 months
  The Modified Barthel Index is a 100-point scale used to assess a patient's proficiency in performing 10 types of Activities of Daily Living (ADL). Each ADL is assigned a numeric value based on the level of assistance the patient requires. Lower scores on the MBI suggest decreased independence, while higher scores indicate greater self-sufficiency. A perfect score of 100 signifies complete independence in basic ADL, whereas the minimum score of 0 indicates total dependence on assistance for these activities. The MBI provides a quantitative measure of an individual's functional status in daily tasks, aiding in the evaluation of their overall independence.

CONTACTS AND LOCATIONS:
Overall Officials: zeest Z hashmi, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Ripah Internationa University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim KH, Jang SH. Effects of Cognitive Sensory Motor Training on Lower Extremity Muscle Strength and Balance in Post Stroke Patients: A Randomized Controlled Study. Clin Pract. 2021 Sep 14;11(3):640-649. doi: 10.3390/clinpract11030079. PMID 34563008
- [Background] Sutcu G, Ozcakar L, Yalcin AI, Kilinc M. BOBATH vs. TASK-ORIENTED TRAINING AFTER STROKE: An assessor-blind randomized controlled trial. Brain Inj. 2023 Jun 7;37(7):581-587. doi: 10.1080/02699052.2023.2203519. Epub 2023 Apr 19. PMID 37074234
- [Background] Ghrouz A, Guillen-Sola A, Morgado-Perez A, Munoz-Redondo E, Ramirez-Fuentes C, Curbelo Pena Y, Duarte E. The effect of a motor relearning on balance and postural control in patients after stroke: An open-label randomized controlled trial. Eur Stroke J. 2024 Jun;9(2):303-311. doi: 10.1177/23969873231220218. Epub 2023 Dec 29. PMID 38158722